CLINICAL TRIAL: NCT01795781
Title: Development of Anticoagulant Assays for New Anticoagulants and Their Reversibility in Vitro
Brief Title: Assays for and Reversal of New Anticoagulants
Status: Completed | Type: Observational
Sponsor: R.P.Herrmann (Other)
Responsible Party: Sponsor-Investigator, R.P.Herrmann, Director, Cell and Tissue Therapies, Western Australia, Royal Perth Hospital
Organization: Royal Perth Hospital (Other)
Other Study IDs: 2011/117
Record Dates: First submitted 2013-02-14; First posted 2013-02-21 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation; Osteoarthritis of the Knee; Osteoarthritis of the Hip
Keywords: Anticoagulant measurement; Anticoagulant reversal; Dabigatran; Rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving a new anticoagulant: Patients are receiving dabigatran for atrial fibrillation or rivaroxaban for osteoarthritis of hip or knee undergoing total hip or knee replacement respectively

SUMMARY:
New anticoagulants are being introduced to replace warfarin. These drugs do not require monitoring and are safer. There is currently no recommended way to reverse these drugs rapidly in the event of undue bleeding or need for emergency surgery. This is a lab study to look at ways to reverse the drugs rapidly

DETAILED DESCRIPTION:
We are developing in vitro assays of measurement of the effect of these drugs on the relevant coagulation pathways in plasma; such assays are not widely established. This will then allow us to test potential reversing agents such as activated Factor VII (Novo-Seven®), or Factor VIII inhibitor bypassing agent (FEIBA) for their ability to reverse these anti-coagulants invitro. The aims of this reversal research strategy is to provide a means whereby patients who present with serious bleeding or who need rapid reversal for surgery, for example, can be offered such treatment to allow rapid normalisation of their coagulation system.

As part of this developmental programme, we wish to obtain samples from patients receiving Rivaroxaban or Dabigatran for therapeutic reasons, to test the effect of the respective drug on the relevant coagulation factors and to test in vitro reversibility.

The only requirement for the patient is to have an extra 20ml of blood taken at a time when the patient is having other blood tests. There are no risks or experimental procedures planned to be carried out on patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving dabigatran for atrial fibrillation
* Or,for osteoarthritis of the hip or knee receiving rivaroxaban to prevent thromboembolic disease after total hip or knee replacement respectively

Exclusion Criteria:

* Failure to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation receiving dabigatran for thrombosis prevention or patients with osteoarthritis of the hip or knee receiving rivaroxaban after total hip or knee replacement respectively for thrombosis prevention
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Ability to reverse anticoagulant effect in vitro of dabigatran or rivarovaban | Two hours after ingestion of anticoagulant dose
  The ability of nonspecific coagulation factors to reverse anticoagulant effect in vitro as measured by dilute thrombin time, Calibrated automated thrombinoscope, thromboelastogram and Rotem

CONTACTS AND LOCATIONS:
Overall Officials: Ross I Baker, MB, BS, Principal Investigator — Royal Perth Hospital, Wellington St, Perth, Australia
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia